CLINICAL TRIAL: NCT00218452
Title: Smoking Cessation for Young Adults Who Binge Drink
Brief Title: Smoking Cessation for Young Adults Who Binge Drink - 1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Ames, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1996-04; R21DA018106 (NIH); R21-18106-1; NIDA-18106-1 (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Adherence; Tobacco Use Cessation; Alcohol & Drug Use; Nicotine Transdermal System
Keywords: Tobacco use cessation
MeSH Terms: conditions — Tobacco Use Cessation; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — assigned to a 6-week individual behavioral treatment involving: 1) a novel brief office intervention for cigarette smoking that includes a treatment component intended to eliminate binge drinking

SUMMARY:
The purpose of this study is develop and test the success of a new smoking cessation intervention that includes a component to eliminate binge drinking.

DETAILED DESCRIPTION:
The primary aim of this pilot investigation is to develop and evaluate the acceptability and feasibility of a novel tobacco dependence intervention that includes a component to eliminate binge drinking. This study will also estimate the magnitude of the effect of the novel intervention on the cigarette smoking behavior of young adult college student smokers.

ELIGIBILITY:
Inclusion Criteria:

(1) Aged 18-25 years. (2) Enrolled as a student at a two or four year technical or non-technical college or university. (3) Smoked > 10 or more cigarettes per day during the past 6 months. (4) Binge drank on > 2 occasions per month during the past 3 months. Binge drinking is defined as consumption of > 5 standardized alcoholic drinks in a row for males or > 4 drinks in a row for females. (5) Able to participate fully in all aspects of the intervention and keep all scheduled appointments. (6) Willing to participate in 6 months of follow-up. (7) Willing to stop smoking and use nicotine patch therapy. (8) Willing to refrain from participating in additional smoking interventions for the duration of the study. (9) Provide written informed consent. (10) General good health as determined by screening physician or registered nurse.

Exclusion Criteria:

(1) Current (past 90 days) alcohol dependence as assessed by the Structured Clinical Interview for DSM-IV Axis I Disorders, Alcohol Dependence Module. (2) Current (past 12 months) non-nicotine or alcohol drug dependence as assessed by a Drug Abuse Screening Test-20 score of > 6. (3) Current elevation of depressive symptoms (past 2 weeks) that would be indicative of clinical depression as assessed by a Beck Depression Inventory-II score of > 20. (4) Current use (past 30 days) of nicotine containing medication or tobacco products other than cigarettes. (5) Current use (past 30 days) of any other smoking cessation treatment involving behavioral or pharmacological interventions. (6) Any medical condition that would preclude use of the nicotine patch including current unstable angina, recent history (past 30 days) of myocardial infarction or stroke, history of severe skin allergies, or evidence of severe chronic dermatosis.

(7) Currently pregnant or breast feeding, or likely to become pregnant during the nicotine patch phase.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Treatment attendance | week 12 and week 24
  quantified as the percentage of sessions attended, will be summarized separately for each treatment group and compared between groups using the rank sum test. One summary will be performed for the percentage of sessions attended face-to-face and a second summary will be performed for the percentage of sessions attended either face-to-face or via telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Ames, Ph.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of North Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota